CLINICAL TRIAL: NCT00516269
Title: A Randomized, Double Blind, Two Period, Placebo-Controlled Crossover Trial of a Sustained Release Methylphenidate in the Treatment of Fatigue in Cancer Patients
Brief Title: Trial of a Sustained Release Methylphenidate in the Treatment of Fatigue in Cancer Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ID00-372
Record Dates: First submitted 2007-08-14; First posted 2007-08-15 (Estimated); Results first posted 2013-04-26 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Breast Cancer; Fatigue; Gastrointestinal Cancer
Keywords: Breast Cancer; Gastrointestinal Cancer; GI Cancer; Fatigue; OROS Methylphenidate HCl; Methylphenidate; Methylphenidate Hydrochloride; Concerta; Ritalin; Placebo
MeSH Terms: conditions — Breast Neoplasms; Fatigue; Gastrointestinal Neoplasms | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Methylphenidate then Placebo (Experimental): Methylphenidate 18 mg oral daily for 2 weeks then Placebo oral daily for 2 weeks
  Interventions: Drug: Methylphenidate; Drug: Placebo
- Placebo then Methylphenidate (Experimental): Placebo oral daily for 2 weeks then Methylphenidate 18 mg oral daily for 2 weeks
  Interventions: Drug: Methylphenidate; Drug: Placebo

INTERVENTIONS:
Drug: Methylphenidate — 18 mg by mouth daily for 2 weeks
  Other Names: Concerta; Ritalin; Methylphenidate Hydrochloride
Drug: Placebo — Capsule by mouth daily for 2 weeks

SUMMARY:
The goal of this clinical research study is to see if the drug OROS Methylphenidate HCl (Concerta) can help to control fatigue in patients with breast, gastrointestinal, lymphoma, myeloma or lung cancer who are going through chemotherapy or hormonal treatment or have completed chemotherapy or hormonal treatment in the last 12 months. The safety of this drug will also be studied. Another goal of the study is to see how certain cytokines change while patients undergo chemotherapy or hormonal treatment.

DETAILED DESCRIPTION:
OROS Methylphenidate HCl is a mild central nervous system stimulant. Cytokines are a type of protein found in blood. Medical researchers here at M. D. Anderson are working to see if they are related to, or can tell us something about, fatigue and its symptoms.

This study will be divided into two, 14-day periods. During one of the 14-day periods, you will be given the study drug. During the other period, you will be given a placebo. A placebo is a sugar tablet that looks just like the study drug tablet.

You will be randomly picked (as in the toss of a coin) to be in one of two treatment groups. In one group you will receive the study drug first and the placebo second. In the other group you receive the placebo first and the study drug second. The chance of being in either treatment group is about equal. Neither you nor the research staff will know which treatment order you are assigned to.

Before treatment starts, you will fill out questionnaires about your level of fatigue, distress, symptoms, and general health. It should take about 5 minutes to complete the questionnaires. You will have a medical history, physical exam (with pulse, temperature, blood pressure), and blood work done. At the start of the study a test of the heart called an EKG will be done. At the start of the study, and after you finish the study, you will complete additional questionnaires that measure mood, fatigue, sleep, and appetite. It should take about 15 minutes to complete the questionnaires. You will also complete a series of tests for memory, visual-motor, and thinking functions. These tests should take about 30 minutes to complete. (This evaluation may take place on or before Day 1 of the study.)

On Day 1, a set of study medications and a diary will be given to you. For the first fourteen days of the study, you will take the assigned study medication (either drug or placebo). Everyday you will fill out the diary, noting the time you took the study medication and answering two questions about your fatigue.

On Day 7, study personnel will see you in the clinic or Ambulatory Treatment Center. The delegated research personnel will take your blood pressure and pulse and ask you about any symptoms or complaints you may have had or any medications you may have taken.

On Day 14, study personnel will see you in the clinic or the Ambulatory Treatment Center where blood pressure and pulse will be measured. Unused study medication will be returned and your diary will be reviewed with the delegated research personnel. You will complete questionnaires asking about fatigue, sleep, depression, and symptoms. It should take about 15 minutes to complete them. You will also complete a series of tests for memory, visual-motor, and thinking functions. The tests should take about 30 minutes to complete. A blood draw will be done to look for changes in hemoglobin and for cytokine analysis.

A new set of study medications and a diary will be given to you. You will follow the same instructions as the first time period. You will take the assigned study medication every morning and fill out the diary, noting the time you took the study medication and answering two questions about your fatigue.

On Day 21, the same activities as Day 7 will occur.

If you are not scheduled to come to M. D. Anderson on Day 7 and Day 21, you will take 2 separate blood pressure measurements 5 minutes apart for each day and report results within 24 hours to the research staff. If you choose to take your blood pressure measurements at home, you need to bring your monitor at study enrollment to have measurements double-checked by research staff.

On Day 28, the study will end. The same activities as Day 14 will occur. In addition, you will have a physical exam.

You will be asked if you prefer the first (first 2 weeks of study) or second (second 2 weeks of study) treatment phase. If you want to continue taking the OROS Methylphenidate you will be allowed to do so off-study as long as there are no medical reasons not to.

This is an investigational study. The study drug has been approved for attention-deficit hyperactivity disorder but is investigational as a treatment for cancer related fatigue. The study medication and physical exams will cost you nothing. You will be reimbursed with a fixed amount of money for each scheduled study visit. The payment will be in the form of a gift card for parking expenses and a gift card for gas expenses. The study doctor or study staff can tell you more about when you will be able to receive reimbursement. A total of 50 patients will take part in this study. All will be enrolled at The University of Texas (UT) MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patient diagnosed with breast, gastrointestinal, lymphoma, myeloma or lung cancer undergoing chemotherapy or hormonal treatment
2. Patient is > or = 18 years of age
3. Patient has Brief Fatigue Inventory "fatigue worst" score of > or = 4 at baseline
4. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status of < or = 2 at baseline
5. Patient has a life expectancy > or = 6 months from the start of the study
6. Patient is using acceptable birth control methods. Female participants (if of child bearing potential and sexually active) and male participants (if sexually active with a partner of child-bearing potential) must use medically acceptable methods of birth control. Medically acceptable methods of contraception include abstinence, birth control pills, diaphragm with spermicide, condom with foam or spermicide, vaginal spermicidal suppository or surgical sterilization
7. Patient must speak and understand English
8. Patient has provided written informed consent to participate in the study prior to enrollment to the study

Exclusion Criteria:

1. History of hypersensitivity reaction to methylphenidate
2. History of or current seizure disorder, glaucoma, major psychiatric diagnosis, narcolepsy, Tourette's syndrome, tension or agitation
3. History of clinically significant cardiac disease.
4. Uncontrolled hypertension: has not been on a stable treatment dose for the past month, or has a systolic pressure consistently (defined as 3 consecutive blood pressure readings within the last 30 days) greater than 150 mm Hg or diastolic pressure consistently greater than 85 mm Hg
5. History of fibromyalgia
6. Use of alcohol while participating in the study
7. Current use of illicit drugs or history of alcohol or drug abuse and/or abuse potential (see protocol for criteria)
8. Moderate to severe depression (> or = 20 on Beck Depression Index II)
9. If taking antidepressants, no changes in dose and/or no start of new course of treatment in the last 30 days
10. Currently taking psychostimulants (including appetite suppressants), monoamine oxidase (MAO) inhibitors, anticoagulant or anticonvulsant therapy
11. Current use of corticosteroids, medications, or stimulants (i.e., vivarin) used to improve fatigue symptoms
12. Use of an investigational medication within the past month
13. Current use of the following herbals or supplements for fatigue relief (DHEA, SAME, ginkgo, ginseng, St. John's Wort (including DHEA, SAME, ginkgo, ginseng, St. John's Wort, metabolite, effedrin, basil, citronella, fennel, horseradish roots, lavender flowers, lemon verbena, marjoram, mint, nettle, pine needles, rosemary, sage, savory, thyme, bay, cayenne pepper, cinnamon, eucalyptus, hyssop, myrrh, oregano, peppermint, ginseng, green, black or Chinese tea, ephedra (aka - ma-huang), popotillo, and Mormon tea)
14. Any coexisting medical condition or are taking any concomitant medication that is likely to interfere with the safe administration of methylphenidate
15. Patients who start epoetin within 30 days prior to enrollment
16. Patients who start taking epoetin during the first week of the study
17. Hemoglobin < 8.0 gm/dl
18. Patients with a thyroid-stimulating hormone (TSH) value > or = 1.5 times the upper limit of normal (ULN)
19. Albumin value 50% lower than the lower limit of normal
20. Evidence of hepatic impairment [total bilirubin > or = 2.5 times ULN (normal range of 0 - 1.0 mg/dl, serum glutamate pyruvate transaminase (SGPT) > or = 2.5 times ULN)]
21. Evidence of renal impairment (serum creatinine > 2.5 times ULN, normal range of 0.8 - 1.5 mg/dl)
22. A severe narrowing (pathological or iatrogenic), obstruction of the gastrointestinal tract, or gastrointestinal malabsorption
23. If taking anxiolytics, and/or hypnotics, no changes in dose and/or no start of new course of treatment in the last 30 days
24. Patients with nausea, vomiting, or diarrhea of Common Toxicity Criteria for Adverse Effects (CTCAE) grade III or higher
25. If taking anticonvulsants for sensory neuropathy (Gabapentin or Pregabalin), no changes in dose and/or no start of new course of treatment in the last 30 days
26. History of severe headaches within 30 days prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2004-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Escalante, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 03/11/2005 to 03/23/2011. All participants were recruited at UT MD Anderson Cancer Center.
Pre-assignment Details: Participants were randomized to receive methylphenidate-placebo or placebo-methylphenidate. Of the 42 enrolled: 33 completed the study + 4 completed partial visits + 1 randomized to placebo twice (38 total), excluded were three who did not meet criteria (not randomized), and one who withdrew consent.
Period: Overall Study
Arm/Group | Methylphenidate Then Placebo | Placebo Then Methylphenidate
Started | 19 | 19
Completed | 17 (2 patients had an early termination) | 16 (2 patients did not complete the study and 1 randomized to placebo twice.)
Not Completed | 2 | 3
Not completed — Adverse Event | 2 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Methylphenidate Then Placebo: 18 mg Oral Daily for 2 Weeks
  Placebo : Capsule By Mouth Daily x 2 Weeks
  Methylphenidate : 18 mg By Mouth Daily x 2 Weeks
- Placebo Then Methylphenidate: Placebo : Capsule By Mouth Daily x 2 Weeks
  Methylphenidate : 18 mg By Mouth Daily x 2 Weeks
- Total: Total of all reporting groups
Arm/Group | Methylphenidate Then Placebo | Placebo Then Methylphenidate | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 19 | 36
  >=65 years | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.26 (11.95) | 51.52 (7.83) | 52.35 (9.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: Mean Difference Between Post-Methylphenidate and Post-Placebo Measurement
Description: The primary endpoint is the "fatigue worst" score (range: 0 - 10) on the Brief Fatigue Inventory (BFI) at the end of two-week treatment (either Methylphenidate or placebo). "Worst fatigue" is defined as participants' rating of worst fatigue on a scale of 0 (no fatigue) to 10 (as bad as can imagine). Since each participant is expected to receive both 2-week of Methylphenidate or 2-week placebo at different times, they serve as their own control. The outcome is the difference in "fatigue worst" score between post-Methylphenidate measurement and post-Placebo measurement.
Time Frame: At end of two 2-week treatment cycles (4 weeks total)
Population: It is a crossover design and only the 33 patients who completed the study were included in the final data analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Methylphenidate: Methylphenidate 18 mg oral daily for 2 Weeks preceded or followed by Placebo oral daily for 2 weeks.
- Placebo: Placebo taken oral daily for 2 Weeks.
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 33 | 33
units on a scale | 5.18 (2.52) | 4.76 (2.68)
Statistical Analysis 1: Comparison: Methylphenidate vs Placebo; As a crossover study, the potential carryover effect was examined first. The pooled data (the 2-week treatment for each intervention i.e. period 1 & period 2) was used to assess the treatment effect (A versus B); Test type: Superiority or Other; p = 0.54, Wilcoxon signed rank test; mean difference in treat versus control = 0.42, Standard Deviation 3.3

ADVERSE EVENTS:
Time Frame: Adverse events were collected for entire study period of 4 weeks.
Arm/Group | Methylphenidate Then Placebo | Placebo Then Methylphenidate
Serious Adverse Events (participants affected / at risk) | 0/19 | 1/19
Other Adverse Events (participants affected / at risk) | 7/19 | 5/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methylphenidate Then Placebo (N=19) | Placebo Then Methylphenidate (N=19)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — The patient was hospitalized for neutropenic fever and was found to have grade 3 anemia. Anemia was not related to the study drug. The SAE is related to chemotherapy administration.
Neutropenic fever (Infections and infestations) | 0 (0) | 1 (1) — One patient was hospitalized for treatment of neutropenic fever. The patient was on the treatment arm. The serious adverse event (SAE) was not related to study drug. The SAE was related to chemotherapy administration for underlying breast cancer.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methylphenidate Then Placebo (N=19) | Placebo Then Methylphenidate (N=19)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nose bleed (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anxiety (Nervous system disorders) | 1 (1) | 0 (0)
Insomnia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Generalized weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination due to slow accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No